CLINICAL TRIAL: NCT02745171
Title: Continuous Behavior Assessment of the Effects of a Physical Therapy Program for Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, MARIA DAS GRAÇAS WANDERLEY DE SALES CORIOLANO, Associate Professor Department of Anatomy at UFPE, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 50967815.7.0000.5208
Record Dates: First submitted 2016-03-30; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Quality of life; Functional mobility; Follow up
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): This group will be evaluated after three months there will be a reassessment, in this case the participating subjects do not perform any kind of therapy.
- Experimental group (Experimental): There will be an initial evaluation, after a month of physical therapy at the end of the protocol, and twice more after the protocol, both interval a month.
  Interventions: Other: physical therapy

INTERVENTIONS:
Other: physical therapy — Will be held 15 sessions, 2 times a week, lasting 50 minutes, a physical therapy protocol developed by the Pro-Parkinson Physiotherapy based on the Guide of the Dutch Society of Physiotherapy (Keus, 2004).
  Arms: Experimental group

SUMMARY:
Introduction: Parkinson's disease (PD) results from dysfunction of the dopaminergic system of degenerative and progressive, with changes in the nigrostriatal pathway, and decreased concentration of dopamine. Has as clinical signs, symptoms called cardinal engines: resting tremor, bradykinesia, rigidity and postural instability. In addition to drug therapy, physical therapy is also considered a useful tool for the treatment of motor disorders of the disease. The role of physiotherapy aims to stimulate the security and independence of patients with PD in carrying out activities and to preserve and improve physical function. Some studies have shown the negative effect of the disease on quality of life and functional mobility. Few studies have been conducted to evaluate the effects of long-term therapy in PD, but many report the beneficial effects of a rehabilitation program in a short period of time.

Objective: To continually assess the effects after the completion of a physical therapy program in patients with Parkinson's disease.

Methods: Type study randomized double blind clinical trial in Parkinson Pro Program Hospital of the Federal University of Pernambuco. Will be recruited subjects with PD, both sexes, in stages 1 to 3 on the scale of Hoehn Yahr and score greater than 18 on the Mini-Mental. Patients who are recruited will undergo an assessment using the scales of assessment of functional mobility, quality of life and motor examination before starting physical therapy at the end of treatment and two months after completion of treatment, and the intervals assessments of a month.

DETAILED DESCRIPTION:
The Parkinson's disease results from dysfunction of the dopaminergic systems, cholinergic, serotonergic and noradrenergic, though the neuropathological basic pattern is the change of the nigrostriatal pathway, with decreased concentration of dopamine at the level of dopamine receptors in the body striatum.

With still little known etiology in most instances, the Parkinson's disease has as clinical signs, symptoms called cardinal engines: resting tremor, bradykinesia, rigidity and postural instability. Additionally, patients may exhibit cognitive deficits and emotional changes with the progression of the disease.

The clinical diagnosis is primarily based on the identification of the cardinal motor symptoms plus the initial response to levodopa therapy . The literature is unanimous in admitting that the use of Levodopa (L-dopa) is the most effective drug for the treatment, and its administration the most recommended in satisfactory symptom control.

In addition to drug therapy, physical therapy is also considered a useful tool for the treatment of motor disorders associated disease. Although the speed of the motor of the patient learningParkinson's disease is lower than their control group of the same age, rehabilitation, these individuals may also acquire motor skills as well as improve their performance through practice repetition.

Although a physical rehabilitation program to be beneficial to improve the activities of daily living (ADL) and mobility in patients with Parkinson's disease , it is not yet clear how long its effect is sustained. Most clinical trials of physiotherapy in PD were based on short-term rehabilitation programs.

Few studies have been conducted to evaluate the effects of long-term physical therapy in Parkinson's disease, but many report the beneficial effects of a short-term rehabilitation program, without having to concern monitoring after the physical therapy.

Thus this study aims to continuously evaluate the behavior of the effects of a physical therapy program in patients with Parkinson's disease.

Knowledge of the time interval which is the decline of the gains from physiotherapy is a guiding point to guide the patient regarding their return to service for revaluation, also considering the fact that the disease have progressive.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Idiopathic Parkinson's disease according to the Bank of London Brain (Hughes et al, 1992);
2. Both sexes;
3. Patients in stages 1 through 3 for this modified version of the Hoehn & Yahr scale (HY);
4. the patient Agreement to participate in the research after explanation and understanding of it and signing the Consent and Informed.

Exclusion Criteria:

1. cognitive disorder identified by the Mini-Mental State Examination as schooling ;
2. Patients with other neurological diseases;
3. initiate other rehabilitative treatment throughout and after the physical therapy program.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
change from quality of life | change in quality of life, it is evaluated every month to complete the four-month period.
  The PDQ-39 is a specific rating scale of QOL in PD and comprises 39 items that can be answered with five different response options: "never"; "On occasion"; "sometimes"; "often"; "Always" or "it is impossible for me."

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886